CLINICAL TRIAL: NCT05458323
Title: Cognitive Level Enhancement Through Vision Exams and Refraction: a Randomized Controlled Trial to Assess Impact of Near and Distance Spectacles on Reducing Rates of Cognitive Decline With Aging in Community Dwelling Older People in India
Brief Title: Cognitive Level Enhancement Through Vision Exams and Refraction
Acronym: CLEVER
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Queen's University, Belfast (Other)
Collaborators: L.V. Prasad Eye Institute (Other); National Institute of Mental Health and Neuro Sciences, India (Other); The George Institute (Other); Johns Hopkins University (Other); University of Michigan (Other); Clearly (Other); Belfast Health and Social Care Trust (Other)
Responsible Party: Principal Investigator, Nathan Congdon, Professor, Queen's University, Belfast
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MHLS 22-13
Record Dates: First submitted 2022-07-11; First posted 2022-07-14 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-12

CONDITIONS: Refractive Errors
Keywords: Cognitive Decline; Elderly; Refractive Error; Spectacles; cost effectiveness analysis; dementia
MeSH Terms: conditions — Refractive Errors; Cognitive Dysfunction; Dementia

STUDY DESIGN:
Intervention Model Description: CLEVER is a single centre, open label, 2-arm, parallel group, stratified, interventional randomised trial, with allocation ratio of 1:1 powered to test superiority of the impact of providing spectacles on rates of cognitive decline among older adults.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Free near and distance glasses (Experimental): All participants randomised to the intervention group will be provided with free near and/or distance spectacles based on the results of refraction. Glasses will be provided at the time of enrolment into the study. The participants will be asked to choose from an assortment of 20 frames. Participants will be asked to report to the study team member in case of any issue with spectacles or if spectacles are lost or broken. Replacement glasses will be provided in case of broken or lost spectacles whenever required. Participants will undergo annual eye exams and refraction, and change of glasses will be prescribed as needed.
  Interventions: Device: Free near and Distance Vision glasses
- Control-No treatment (No Intervention): All participants randomised to the control group will receive a prescription for spectacles and given free near and/or distance glasses as needed at study close out.

INTERVENTIONS:
Device: Free near and Distance Vision glasses — Intervention Description: All participants randomised to the intervention group will be provided with free near and/or distance spectacles based on the results of refraction.Glasses will be provided at the time of enrolment in the study.
  Arms: Free near and distance glasses

SUMMARY:
The investigators aim to conduct a mixed-method study in which a randomised controlled trial (RCT) and a descriptive qualitative study will be conducted. The RCT aims to determine whether free near and distance glasses provided to residents in Hyderabad, India, aged ≥ 60 years, with under- or un- corrected refractive error and normal baseline hearing and cognition (HMSE > 18), can improve quality of life, reduce falls, reduce depression, improve social interaction and physical activity cost-effectively over 36 months. The primary qualitative research aim is to a) contextualize the RCT with information on the milieu and culture in which the trial will be conducted; b) provide data on the lived experiences of older adults with reduced vision in the study area, and c) conduct a process evaluation of the trial.

The primary outcome measure is the three-year change in cognition measured by LASI- DAD (Longitudinal Aging Study in India(LASI)- Diagnostic Assessment of Dementia(DAD) global cognitive score.

Secondary Outcome Measures: Three year change in Quality of Life score measured by WHO QOL-BREF; Visual functioning from the RASCH-scaled version of INDVFQ(Indian Visual Functioning(INDVFQ);self-reported physical activity score measured using IPAQ questionnaire; PHQ9 score; domain specific cognitive score (orientation, executive function, language/fluency, memory) measured by HMSE; Total cost of care including direct and indirect costs; Quality adjusted life years; Incremental Cost Effectiveness Ratio; Number of falls measured by Quick Screen score over the three years; Social network density at 3 years (SNI 1-3 represents a "limited" social network, 4-5 is a "medium" social network, and SNI ≥6 is a "diverse" social network) measured by the SNI score; An additional secondary outcome will be LASI-DAD global cognitive score analysed by excluding any tests determined pre-hoc to depend on visual acuity.

DETAILED DESCRIPTION:
The number of people living with dementia globally will rise from 50 million in 2017 to 131.5 million by 2050. The majority reside in low and middle-income countries (LMICs), where a 223% increase in the burden of dementia is expected from 2015 to 2050. The household cost of caring for demented relatives in India was £2.48 billion in 2013, where total expenses for dementia care will soon consume 0.5% of Gross Domestic Product (GDP). Despite the rapidly-growing burden of dementia in India, only 1 in 10 affected are diagnosed or treated. Proven preventive strategies are desperately needed to close the gap, and could reduce incidence by an estimated 41%, especially early, at the stage of mild cognitive impairment, which itself increases risk of dementia by 23-fold. Existing interventions have predominantly been evaluated in high-income countries (HIC), despite the acknowledged need for prevention in low resource settings. India's national dementia strategy, documented in the Alzheimer's and Related Society of India (ARDSI) Report (2018) and Dementia in India (2020), echo the WHO Dementia Global Action Plan (2017) in prioritising evidence-based approaches to reduce risk.

The elderly, at greatest risk for cognitive disorders, also have the highest prevalence of vision impairment, which affects 2.2 billion persons globally. Growing longitudinal evidence links vision impairment and risk of cognitive decline, with population studies in the United States reporting a 55% increased 9-year risk of new cognitive impairment among visually impaired persons. Longitudinal studies elsewhere in the United States, France, Singapore and China report similar results. While vision impairment is a strong predictor of future cognitive performance, cognition is relatively weakly linked to future visual decline. Both distance impairment and impairment of near vision, a nearly universal part of aging without refractive correction, have been implicated. Observational studies also suggest vision care slows rates of cognitive decline by up to 50%. The association between vision loss and cognitive decline and dementia, while consistent and strong, is not well understood, and various causal pathways have been posited. These include common neurodegenerative or micro vascular aetiology, increased cognitive load, and limited social contact and physical activity due to poor vision, each independently shown to elevate risk of dementia. Studies investigating the role of vision correction in slowing cognitive decline will have a significant impact in developing strategies to reduce the burden of dementia.

Design: single centre, open label, two-arm, parallel group, stratified, interventional randomised trial with a qualitative component Rationale: Despite considerable longitudinal observational evidence, there have been no randomised trials to investigate whether providing near and distance glasses can slow cognitive decline in the elderly. Proof of a causative association between vision correction and the slowing of cognitive decline is needed to potentiate investment in inexpensive vision care for prevention. This requires randomised trials, and none have yet been done.

Study Plan:

Eligibility assessments conducted for 5000-10000 participants. After providing the consent and meeting the eligibility criteria, 820 participants randomised to intervention and control groups.

HbA1C and information about oral health will be collected from the participants in the follow-up visits.

Annual follow-ups for 3 years for both groups. Cataract follow up: Along with annual visits and the spectacle compliance contacts, follow-up would also be done for those participants who are advised for cataract surgery and efforts would be made to ensure they get the cataract surgery done. This surgery would be done at no cost to the patient.

Lost to follow ups documented with reason for both groups. Missed data for both groups will be analysed as intention to treat (ITT) analysis.

Statistical methods: The change in LASI-DAD global cognitive score between baseline and 36 months will be compared between the intervention and control groups. A linear mixed model will be used to estimate the overall change in LASI-DAD global cognitive score over-time adjusting for potential determinants of change in cognitive status, such as baseline cognitive score, age, gender, education level, occupation, quality of life, depression, social interaction, and physical activity. Restricted maximum likelihood estimation (REML) will be used as the estimation method. If the LASI-DAD global cognitive score is skewed, the log transformation will be used and if the data contains zero, the square root transformations will be done (since the log of zero is undefined). The log transformation is mainly preferred for its ease use and interpretability. The mean change score (and its 95% CI) will be reported for 12 months versus baseline and 24 months versus baseline, and 36 months versus baseline. Significance tests will be two-sided with 5% level of significance and reported using overall Wald p-values for linear regression. All continuous outcomes (INDVFQ, IPAQ, PHQ9, HMSE scores) will be analysed following the same procedure as the main outcome. SNI (categorical ) will be analysed using the multinomial logistic regression. Further details will be provided in the SAP

The trial anticipates two intercurrent events: (i) cataract surgery and (ii) cataract development with refusal of surgery. The primary estimand uses a treatment policy strategy including all patients regardless of cataract status or surgery. The secondary estimand uses a treatment policy for surgery and a hypothetical strategy for refusal, censoring at refusal.

Justification for sample size: Imputing three-year un-intervened decline in the outcome variable (LASI-DAD global score from cross-sectional, age-stratified data, at 29% effect size (from the ACHIEVE study), 502 participants give 90% power at p = 0.05 (two-tailed) based on a two-sample test. With annual follow-up loss of 13% based on estimation from previous studies conducted in India and WHO annual mortality rates in the elderly Indian population (ranging between 10.1 % and 12.7 %) a total of 760 participants is required.

To align with the estimands framework, and to account for intercurrent events that may impact outcome assessment (e.g. loss to follow-up, the development of cataract or competing risks), the sample size was further adjusted. Assuming 7% missing data for the intercurrent events and using the formula by Fang and Jin (2021), 820 total participants are needed across the two study groups. This ensures appropriate power for the primary analysis under a missing-at-random assumption.

With 60% prevalence of uncorrected distance and/or near refractive error, the total number of people needing to be screened is estimated at approximately 1370. However, based on available and other local factors as evident from pre-pilot work, 5,000-10,000 participants may have to be screened for recruiting 820 participants for the trial.

ELIGIBILITY:
Inclusion Criteria

1. Community dwelling
2. Residency

   a. Participants must plan to reside in the local area for the study duration
3. Presenting vision in the better eye due to uncorrected refractive error

   1. Impaired distance vision less than 6/18
   2. Near vision less than N6 at 40 cm
4. Willingness

   1. to participate
   2. to be randomized
   3. to adhere to the protocol

Exclusion criteria

1. Impaired baseline cognition

   a. HMSE score less than or equal to 18
2. Non-refractive causes of vision impairment
3. Severely impaired mobility

   1. immobile
   2. bedridden
   3. wheelchair
   4. using walker
4. Severe medical illness likely to limit the life span

   1. Cancer
   2. Heart disease
   3. Stroke
   4. HIV or AIDS
   5. Chronic lung disease
   6. Kidney disease
5. Hearing loss assessment

   1. self-reported hearing impairment
   2. inability to hear
   3. fail in whisper test hearing screening(unable to repeat three out of six words)

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 820 (Estimated)
Dates: Start 2024-01-18 (Actual); Primary Completion 2027-11-30 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in cognitive score | Time point(s) of primary interest: 36 months collected at 12, 24 and 36 months
  The metric or method of measurement to be used: LASI-DAD global cognitive score. The best possible score is 360 and the worst possible score is 0.

SECONDARY OUTCOMES:
26-Item Quality of Life | Time point(s) of primary interest: 36 months collected every 12 months - ie at 12, 24 and 36 months
  The metric or method of measurement to be used: Quality of Life using WHO BREF questionnaire. Higher scores (for 4 domains) indicate higher quality of life and vice versa (it is a continuum)
Cost effectiveness | Time point(s) of primary interest: 36 months collected every 12 months - ie at 12, 24 and 36 months
  The metric or method of measurement to be used: Cost-effectiveness using Client Service Receipt Inventory
Social interaction/isolation | Time point(s) of primary interest: 36 months collected every 12 months - ie at 12, 24 and 36 months
  The metric or method of measurement to be used: Social Networking Index. The best possible score is 12 and the worst possible score is 0
Self-reported physical activity. | Time point(s) of primary interest: 36 months collected every 12 months - ie at 12, 24 and 36 months
  The metric or method of measurement to be used: International Physical Activity Questionnaire Self-reported physical activity: International Physical Activity Questionnaire (IPAQ).
Falls | Time point(s) of primary interest: 36 months collected every 12 months - ie at 12, 24 and 36 months
  The metric or method of measurement to be used: Quick Screen for falls Risk. The worst possible score is 7% and the best possible score is 49%
Depression | Time point(s) of primary interest: 36 months collected every 12 months - ie at 12, 24 and 36 months
  The metric or method of measurement to be used: Patient Health Questionnaire, PHQ9. Worst score is 0 and best possible score is 27
Glasses compliance | Time point(s) of primary interest: 36 months collected every 12 months - ie at 12, 24 and 36 months
  The metric or method of measurement to be used: Use of glasses during follow-up visits. The best possible score is 1 and the worst possible score is 0
Visual Function | Time point(s) of primary interest: 36 months collected every 12 months - ie at 12, 24 and 36 months
  The metric or method of measurement to be used: Indian VFQ. The measure will be in logits (using Rasch-scaled interval scores) and it is a continuum with positive person scores indicating lower visual functioning and negative scores indicating better visual functioning.
Domain-specific cognitive function | Time point(s) of primary interest: 36 months collected every 12 months - ie at 12, 24 and 36 months
  The metric or method of measurement to be used: Hindi Mental State Examination. The best possible score is 31 and the worst possible score is 0.

CONTACTS AND LOCATIONS:
Overall Officials: Nathan G Congdon, MD, MPH, Principal Investigator — Queen's University, Belfast; Rohit C Khanna, MPH, Principal Investigator — L.V. Prasad Eye Institute; Suvarna Alladi, DM, Principal Investigator — National Institute of Mental Health and Neuro Sciences, India
Locations (1):
- L V Prasad Eye Institute, Hyderabad, Telangana, India

IPD SHARING:
Plan to Share IPD: Yes
All Individual Participant Data(IPD) will be stored in anonymised format. The IPD that includes personal identifiable information will be deleted when the data collection process is complete and before the initiation of data analysis.
  Only de-identified data will be shared with all the researchers for analysis. The primary analysis will be conducted on all outcome data obtained from all enrolled participants as randomised.
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: All deidentified IPD will be available from September 2022 (anticipated Trial start date) to September 2035 (inclusive of analysis, publication and archival).
Access Criteria: Following publication of the primary and secondary outcomes there may be scope to conduct additional analyses on the data collected. In such instances formal requests for data will need to be made in writing to the Chief Investigator, who will discuss this with the Sponsor. The study will comply with the good practice principles for sharing individual participant data from publicly funded clinical trials and data sharing will be undertaken in accordance with the required regulatory requirements

REFERENCES:
- [Result] Marmamula S, Alladi S, Umapathy K, Chan VF, MacKenzie G, Lohfeld L, Mettla AL, Rayasam S, Gothwal VK, Narayanan R, Pyda G, Chadalavada HP, Thomas P, Sigwadhi LN, Azuara-Blanco A, McDowell C, McMullan S, Murphy L, Clarke M, Ehrlich JR, Sweenor B, O'Neill C, Komaravolu S, Maulik PK, Murthy GVS, Kumar K, Nyshadham A, Adhvaryu A, McCabe C, Bloom DE, Lee J, Lin F, Coghlan S, Khanna RC, Congdon N. Cognitive Level Enhancement through Vision Exams and Refraction (CLEVER): study protocol for a randomised controlled trial. Trials. 2025 Mar 28;26(1):109. doi: 10.1186/s13063-025-08813-x. PMID 40156032